CLINICAL TRIAL: NCT05091359
Title: Unstable Proximal Femur Transtrochanteric Fractures Treated With Dynamic Hip Screw and ß -Tricalcium Phosphate/ Hemihydrated Calcium Sulfate Graft Scaffold
Brief Title: Femur Transtrochanteric Fractures Treated With Dynamic Hip Screw and Calcium Sulfate Scaffold.
Acronym: geneX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Regional Tlalnepantla (Other Government)
Responsible Party: Principal Investigator, Julio Carlos Velez de Lachica, Md. High Specialty Associate Professor of the Joint Surgery Course, Hospital Regional Tlalnepantla
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 02
Record Dates: First submitted 2021-09-03; First posted 2021-10-25 (Actual); Last update posted 2021-10-25 (Actual); Status verified 2021-10

CONDITIONS: Proximal Femur Fracture
Keywords: Dynamic Hip Screw; DHS HIP FRACTURE
MeSH Terms: conditions — Proximal Femoral Fractures

STUDY DESIGN:
Intervention Model Description: A two group comparison
Who Masked: Participant
Masking Description: The procedure was elected by participant randomization.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Experimental): Participants in which absorbable graft of tricalcium ß phosphate / calcium sulfate hemihydrate paste at the time of the placement of the hip implant to prevent loosening of it's unstable trans-trochanteric fractures of the proximal femur, were applied.
  Interventions: Device: Study group with absorbable graft of tricalcium ß phosphate / calcium sulfate hemihydrate paste
- Control Group (No Intervention): Participants without application of graft during hip implant.

INTERVENTIONS:
Device: Study group with absorbable graft of tricalcium ß phosphate / calcium sulfate hemihydrate paste — Application of absorbable graft of tricalcium ß phosphate / calcium sulfate hemihydrate in paste for prevent loosening of Dynamic Hip Screw implant
  Arms: Study group

SUMMARY:
This is a randomised prospective comparison study to evaluate the incidence of cut - out failure of the dynamic hip screw implant alone compared to the dynamic hip screw adding calcium sulfate through the cervical canal before placing the sliding screw for improvement of the implant stability integration and bone healing.

DETAILED DESCRIPTION:
Transtrochanteric fractures are a frequent entity, mainly in patients over 65 years old, with low bone density. Most of these fractures of the proximal femur are treated effectively with internal fixation with dynamic hip screw (DHS), nonetheless a conditional factor in the treatment success its in the fracture stability and in the osteoporosis severity.

There is controversy in the treatment decision in patients with osteoporosis and an unstable fracture added the risk of peri-prosthetic infection or increased bleeding during surgery means that the decision to place a DHS versus a prosthesis is debated.

This study represents the first comparison of closed reduction and internal fixation with DHS using calcium sulfate graft versus conventional DHS procedure.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 65 and 80 years old
* Patients classified as 31A1.3 and all 31A2 by the Orthopaedic Trauma Association classification system.

Exclusion Criteria:

* Patients with stable hip fractures
* Participants who do not accept the randomization process
* patients who do not complete follow-up during the study

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 36 (Actual)
Dates: Start 2015-04-01 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2019-05-10 (Actual)

PRIMARY OUTCOMES:
Incidence of cut - out failure of the dynamic hip screw implant in unstable transtrochanteric fractures | 12 weeks for each patient
  The aim of this study is to evaluate the incidence of cut - out failure of the dynamic hip screw implant alone compared to the dynamic hip screw adding calcium sulfate through the cervical canal before placing the sliding screw to improve implant integration and bone healing.

CONTACTS AND LOCATIONS:
Overall Officials: JULIO C VELEZ, mD, Principal Investigator — HEAD OF THE ORTHOPEDIC SERVICE OF THE REGIONAL HOSPITAL TLALNEPANTLA ISSEMYM; SILVIA S SERRANO REYES, MD, Study Chair — JOINT SURGERY RESIDENT

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hassankhani EG, Omidi-Kashani F, Hajitaghi H, Hassankhani GG. How to Treat the Complex Unstable Intertrochanteric Fractures in Elderly Patients? DHS or Arthroplasty. Arch Bone Jt Surg. 2014 Sep;2(3):174-9. Epub 2014 Sep 15. PMID 25386578
- [Background] Brox WT, Roberts KC, Taksali S, Wright DG, Wixted JJ, Tubb CC, Patt JC, Templeton KJ, Dickman E, Adler RA, Macaulay WB, Jackman JM, Annaswamy T, Adelman AM, Hawthorne CG, Olson SA, Mendelson DA, LeBoff MS, Camacho PA, Jevsevar D, Shea KG, Bozic KJ, Shaffer W, Cummins D, Murray JN, Donnelly P, Shores P, Woznica A, Martinez Y, Boone C, Gross L, Sevarino K. The American Academy of Orthopaedic Surgeons Evidence-Based Guideline on Management of Hip Fractures in the Elderly. J Bone Joint Surg Am. 2015 Jul 15;97(14):1196-9. doi: 10.2106/JBJS.O.00229. No abstract available. PMID 26178894
- [Background] Quinn RH, Mooar PA, Murray JN, Pezold R, Sevarino KS. Treatment of Hip Fractures in the Elderly. J Am Acad Orthop Surg. 2017 May;25(5):e102-e104. doi: 10.5435/JAAOS-D-16-00431. PMID 28379914
- [Background] Singh S, Shrivastava C, Kumar S. Hemi replacement arthroplasty for unstable inter-trochanteric fractures of femur. J Clin Diagn Res. 2014 Oct;8(10):LC01-4. doi: 10.7860/JCDR/2014/10171.4972. Epub 2014 Oct 20. PMID 25478376
- [Background] Kim Y, Moon JK, Hwang KT, Choi IY, Kim YH. Cementless bipolar hemiarthroplasty for unstable intertrochanteric fractures in octogenarians. Acta Orthop Traumatol Turc. 2014;48(4):424-30. doi: 10.3944/AOTT.2014.13.0119. PMID 25230266
- [Background] Swart E, Makhni EC, Macaulay W, Rosenwasser MP, Bozic KJ. Cost-effectiveness analysis of fixation options for intertrochanteric hip fractures. J Bone Joint Surg Am. 2014 Oct 1;96(19):1612-20. doi: 10.2106/JBJS.M.00603. PMID 25274786
- [Background] Kregor PJ, Obremskey WT, Kreder HJ, Swiontkowski MF. Unstable pertrochanteric femoral fractures. J Orthop Trauma. 2014 Aug;28 Suppl 8:S25-8. doi: 10.1097/BOT.0000000000000187. PMID 25046412
- [Background] De Bruijn K, den Hartog D, Tuinebreijer W, Roukema G. Reliability of predictors for screw cutout in intertrochanteric hip fractures. J Bone Joint Surg Am. 2012 Jul 18;94(14):1266-72. doi: 10.2106/JBJS.K.00357. PMID 22810396
- [Background] Hsueh KK, Fang CK, Chen CM, Su YP, Wu HF, Chiu FY. Risk factors in cutout of sliding hip screw in intertrochanteric fractures: an evaluation of 937 patients. Int Orthop. 2010 Dec;34(8):1273-6. doi: 10.1007/s00264-009-0866-2. Epub 2009 Sep 26. PMID 19784649
- [Background] Wu CC, Shih CH, Chen WJ, Tai CL. Treatment of cutout of a lag screw of a dynamic hip screw in an intertrochanteric fracture. Arch Orthop Trauma Surg. 1998;117(4-5):193-6. doi: 10.1007/s004020050228. PMID 9581243
- [Background] Puram C, Pradhan C, Patil A, Sodhai V, Sancheti P, Shyam A. Outcomes of dynamic hip screw augmented with trochanteric wiring for treatment of unstable type A2 intertrochanteric femur fractures. Injury. 2017 Aug;48 Suppl 2:S72-S77. doi: 10.1016/S0020-1383(17)30498-9. PMID 28802425
- [Background] Valentini R, Martino M, Piovan G, De Fabrizio G, Fancellu G. Proximal cut-out in pertrochanteric femural fracture. Acta Biomed. 2014 Aug 20;85(2):144-51. PMID 25245650

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2020-10-03): https://cdn.clinicaltrials.gov/large-docs/59/NCT05091359/Prot_SAP_ICF_000.pdf